CLINICAL TRIAL: NCT03237221
Title: Clinical Characteristics, Treatment and Prognosis of Chest Tightness Variant Asthma
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, yanfugui, Vice Director，Respiratory and Critical Care Medicine，Clinical Vice Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: CTVA-China
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Chest Syndrome; Clinical Anxiety; Clinical Depression; Lung Function; Quality of Life; Eosinophilia; Nitric Oxide; Airway Responsiveness; Induced Sputum
MeSH Terms: conditions — Asthma; Depressive Disorder, Major; Eosinophilia | interventions — Guidelines as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Treat patient according to Global Initiative for Asthma (GINA) guideline — Treat patient according to Global Initiative for Asthma (GINA) guideline

SUMMARY:
Asthma, abbreviation for bronchial asthma, is one of the common chronic airways disease that threatens human health. Typical symptoms of asthma are recurrent wheezing, shortness of breath, chest tightness and cough, usually occurring at night or early morning. However, there are still some patients with only persistent clinical manifestations of chest tightness. Concerned about this group of patients, we presented a subgroup of bronchial asthma, namely, chest tightness variant asthma (CTVA). This asthma subgroup usually lacks asthma-specific clinical features such as wheezing, shortness of breath, wheezing, and therefore often misdiagnosed for a long time. In order to further understand the clinical characteristics, pathogenesis, and prognosis of patients with CTVA, we conducted a national multicenter observation study to further understand CTVA. Finally, we plan to clarify whether CTVA is a relatively independent asthma phenotype. Meanwhile, reducing misdiagnosis and perform an appropriate treatment of CTVA.

ELIGIBILITY:
Inclusion Criteria:

1. all subjects agreed to participate, understand the project, observe the use of drugs, agree to follow-up, and signed informed consent;
2. the age of more than 14 and less 80 years old, gender and ethnicity are not limited;
3. the duration time was more than 6 months,and chest tightness was the only complaint, without breathing, short of breath, chronic cough;
4. no wheezing;
5. a diagnosis of asthma supported by one or more other characteristics:

   * bronchial provocation test positive;
   * improvement in forced expiratory volume at one second (FEV1) of more than 12% and 200 mL after inhaled salbutamol;
   * variability in diurnal peak expiratory flow (PEF) of more than 10% for one day during one week.
6. bronchodilator and glucocorticoid treatment is effective;
7. exclude the following diseases by the corresponding doctors: coronary heart disease, myocarditis, heart failure, GERD, neuromuscular disease, and mental disease.

Exclusion Criteria:

1. can not cooperate with related inspection or for other reasons;
2. patients with chronic obstructive pulmonary disease, interstitial pneumonia, active tuberculosis, community acquired pneumonia, lung cancer, bronchiectasis, cor pulmonale, pulmonary embolism, and accompanied with serious systematic disease (such as coronary heart disease, myocarditis, heart failure, gastroesophageal reflux disease, neuromuscular disease, etc);
3. history of drug abuse, alcohol abuse or anesthesia or with a history of mental illness (schizophrenia, obsessive-compulsive disorder, depression) and against personality, motivation, suspicious, or other emotional or mental issues that may affect participation in the study;
4. taking part in other drug clinical trial project, or drop out less than 3 months;
5. during pregnancy, lactation women;
6. obvious abnormal of High Resolution CT.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with only symptom of chest tightness and bronchial provocation test positive according to eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Asthma control questionnaire (ACQ) | Change from Baseline ACQ score at 36 months
  Asthma control questionnaire (ACQ)

SECONDARY OUTCOMES:
Forced expiratory volume in one second | Change from Baseline ACQ score at 36 months
  Forced expiratory volume in one second
Airway responsiveness | Change from Baseline ACQ score at 36 months
  Airway responsiveness
Peak expiratory flow | Change from Baseline ACQ score at 36 months
  Peak expiratory flow
Asthma quality of life questionnaire | Change from Baseline ACQ score at 36 months
  Asthma quality of life questionnaire
Acute asthma episode | Change from Baseline ACQ score at 36 months
  Acute asthma episode
Numbers of emergency or hospitalization | Change from Baseline ACQ score at 36 months
  Numbers of emergency or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Huahao Shen, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (34):
- China (34):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital，Third Military Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital，Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital, Nanfang Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital,Guangzhou Medical University, Guangzhou, Guangdong
  - People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Affiliated Hospital,Zhanjiang Medical College, Zhanjiang, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Central Hospital of Shenyang Military, Shenyang, Liaoning
  - The First Affiliated Hospital, China Medical University, Shenyang, Liaoning
  - Xijing Hospital, Xi'an, Shaanxi
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Shandong Provincal Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Weifang Asthma Hospital, Weifang, Shandong
  - Yantai liuhuanding Hospital, Yantai, Shandong
  - Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality
  - No.1 Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Tongji Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw hospital, College of Medicine，Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The Second Affiliated Hospital,Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided